CLINICAL TRIAL: NCT04286308
Title: Cortical-Basal Ganglia Speech Networks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert Mark Richardson, Director of Functional Neurosurgery, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019P003841
Record Dates: First submitted 2020-01-08; First posted 2020-02-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease; Essential Tremor; Dystonia
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain signal data collection (Experimental): Brain signal data collection at the time of deep brain stimulation (DBS) surgery.
  Interventions: Other: electrophysiological data collection

INTERVENTIONS:
Other: electrophysiological data collection — Electrophysiological data collection at the time of DBS surgery.

SUMMARY:
In this research study the researchers want to learn more about brain activity related to speech perception and production.

DETAILED DESCRIPTION:
Speech production is disrupted in a number of neurological diseases that involve the basal ganglia, including Parkinson's disease (PD) and dystonia. The investigators will use a novel experimental approach and combination of analytic techniques to elucidate the contribution of neural activity in cortical-basal ganglia circuits to the hierarchical control of speech production, in subjects undergoing deep brain stimulation surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled for DBS implantation, as determined by the clinical multidisciplinary movement disorders board with definitive diagnosis of Parkinson's disease, essential tremor or dystonia.
2. Subjects able to provide informed consent and comply with task instructions.
3. Subjects 18-85 years old

Exclusion Criteria:

1. Subjects with reported hearing loss.
2. Non-English-speaking subjects

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The number of subjects providing the interpretable speech related electrophysiological data collection. | Duration of single DBS surgery
  The number of subjects providing the interpretable speech related electrophysiological data during DBS surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No